CLINICAL TRIAL: NCT00724568
Title: A Multi-Institutional Phase I/II Study of Revlimid® (Lenalidomide), Velcade® (Bortezomib), Dexamethasone, and Doxil®, (RVDD) Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Combination Study of Revlimid®, Velcade® Dexamethasone and Doxil® (RVDD)for Newly Diagnosed Multiple Myeloma
Acronym: RVDD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.098; HUM 12962 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2008-04-11; First posted 2008-07-29 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Drug Therapy (Experimental): Patients will be treated with Velcade at 1.3 mg/m2 on days 1, 4, 8, and 11, Doxil at indicated doses on day 4, Dexamethasone at 20 mg orally on days of Velcade and the day after for all dose levels, and Revlimid at indicated doses on days 1-14 in 3-week cycles for 4-8 cycles. To determine the MTD of the combination of Revlimid, Velcade, dexamethasone, and Doxil, four dose levels are planned.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Doxil

INTERVENTIONS:
Drug: Lenalidomide — Patients will be treated with Revlimid on days 1-14 in 3-week cycles for 4-8 cycles.
  Other Names: Revlimid
Drug: Bortezomib — Patients will be treated with Velcade at 1.3 mg/m2 on days 1, 4, 8, and 11
  Other Names: Velcade
Drug: Dexamethasone — Patients will be treated with Dexamethasone at 20 mg orally on days of Velcade and the day after for all dose levels.
Drug: Doxil — Patients will be treated with Doxil on day 4.

SUMMARY:
This research study is evaluating an investigational combination of four drugs called Revlimid® (lenalidomide), Velcade® (bortezomib), Dexamethasone and Doxil® (RVDD) as a possible treatment for newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
During the Phase I portion of this clinical trial, the doses of Revlimid® and Doxil® will be increased until the best and safest amount (or dose) is identified in combination with Velcade® and Dexamethasone. "Investigational" means that the drug combination is still being studied and that research doctors are trying to find out more about it such as the safest dose to use, the side effects it may cause and how effective the Velcade®, Doxil®, Dexamethasone and Revlimid® investigational combination is for treating newly diagnosed multiple myeloma. In this clinical trial we are looking for the highest dose of the combination that can be given safely and see how well it works as a combination in newly diagnosed patients.

Each of these drugs, Velcade®, Doxil®, Dexamethasone and Revlimid® are approved by the FDA (U.S. Food and Drug Administration). They have not been approved in this combination for use for your type of cancer or any other type of cancer. Velcade® is currently approved by the United States Food and Drug Administration (US FDA) for the treatment of multiple myeloma patients who have received at least one prior therapy. Doxil® has recently been approved by the US FDA for multiple myeloma in combination with Velcade® in patients who have not previously received Velcade® and have received at least one prior therapy. Dexamethasone is commonly used, either alone, or in combination with other drugs, to treat multiple myeloma. Revlimid® is currently approved by the US FDA in combination with dexamethasone for the treatment of patients with multiple myeloma who have received at least 1 prior therapy.

After the Phase I clinical trial defines the safest doses of Velcade®, Doxil®, Dexamethasone and Revlimid® that can be taken together, the research study will move on to its second portion, a Phase II clinical trial. The Phase II portion of the clinical trial will test the clinical effectiveness of the best dose combination of the four drugs.

ELIGIBILITY:
Inclusion Criteria

* At least 18 years of age at the time of consent
* Measurable disease
* All necessary baseline studies completed
* LVEF (left ventricular ejection fraction) greater than or equal to 50 percent by MUGA (multigated acquisition scan) or ECHO (echocardiogram)
* Must be able to adhere to study visit schedule

Exclusion

* Greater than or equal to grade 2 peripheral neuropathy on clinical examination within 14 days of enrollment
* Renal insufficiency
* Evidence of mucosal or internal bleeding and/ or platelet refractory.
* Absolute neutrophil count less than 1000 cells/mm^2 within 14 days of enrollment.
* Acceptable labs
* Concomitant medications that include corticosteroids
* Myocardial infarction within 6 months prior to enrollment, uncontrolled angina, severe uncontrolled ventricular arrhythmias
* Clinically relevant active infection or serious medical condition that places the subject at unacceptable risk
* Any condition, including laboratory values that places the subject at an unacceptable risk
* Another malignancy within 3 years of enrollment, with the exception of the complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy
* Hypersensitivity to bortezomib, boron, or mannitol or any of the components of DOXIL
* Female subject that is pregnant or breastfeeding.
* Can not have received any other investigational drugs within 14 days of enrollment
* Serious medical or psychiatric illness
* Uncontrolled diabetes mellitus
* Hypersensitivity to acyclovir or similar antiviral drug
* POEMS (plasma cell dyscrasia with polyneuropathy)
* Known HIV
* Known hepatitis B or C
* Known intolerance to steroid therapy
* Known hypersensitivity to required prophylactic mediations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2014-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Talpaz, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (6):
- United States (5):
  - Emory University Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute (and Massachusetts General), Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - The Ohio State University Medical Center, Columbus, Ohio
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Jakubowiak AJ, Griffith KA, Reece DE, Hofmeister CC, Lonial S, Zimmerman TM, Campagnaro EL, Schlossman RL, Laubach JP, Raje NS, Anderson T, Mietzel MA, Harvey CK, Wear SM, Barrickman JC, Tendler CL, Esseltine DL, Kelley SL, Kaminski MS, Anderson KC, Richardson PG. Lenalidomide, bortezomib, pegylated liposomal doxorubicin, and dexamethasone in newly diagnosed multiple myeloma: a phase 1/2 Multiple Myeloma Research Consortium trial. Blood. 2011 Jul 21;118(3):535-43. doi: 10.1182/blood-2011-02-334755. Epub 2011 May 19. PMID 21596852

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I; Phase II: Patients will be treated with Velcade at 1.3 mg/m2 on days 1, 4, 8, and 11, Doxil at indicated doses on day 4, Dexamethasone at 20 mg orally on days of Velcade and the day after for all dose levels, and Revlimid at indicated doses on days 1-14 in 3-week cycles for 4-8 cycles.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 42 | 32
Completed | 42 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 74 patients were enrolled in this phase 1/2 study. 2 patients were not evaluable for the Dose Limiting Toxicity (DLT) and therefore only 72 are included in the baseline analysis population.
Groups:
- Combination Drug Therapy: Patients will be treated with Velcade at 1.3 mg/m2 on days 1, 4, 8, and 11, Doxil at indicated doses on day 4, Dexamethasone at 20 mg orally on days of Velcade and the day after for all dose levels, and Revlimid at indicated doses on days 1-14 in 3-week cycles for 4-8 cycles.
Arm/Group | Combination Drug Therapy
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Combination Therapy With VELCADE, Dexamethasone, and Doxil, (RVDD)
Description: Dose Level 1:
  15 mg Revlimid daily on days 1-14 followed by 7-day rest every 21 days 1.3 mg/m2 Velcade daily on days 1, 4, 8 and 11 20 mg dexamethasone daily on Days 1, 2, 4, 5, 8, 9, 11, 12* and 20 mg/m2 Doxil daily on day 4
  Dose Level 2:
  20 mg Revlimid daily on days 1-14 followed by 7-day rest every 21 days 1.3 mg/m2 Velcade daily on days 1, 4, 8 and 11 20 mg dexamethasone daily on Days 1, 2, 4, 5, 8, 9, 11, 12* and 20 mg/m2 Doxil daily on day 4
  Dose Level 3:
  25 mg Revlimid daily on days 1-14 followed by 7-day rest every 21 days 1.3 mg/m2 Velcade daily on days 1, 4, 8 and 11 20 mg dexamethasone daily on Days 1, 2, 4, 5, 8, 9, 11, 12* and 20 mg/m2 Doxil daily on day 4
  Dose Level 4:
  25 mg Revlimid daily on days 1-14 followed by 7-day rest every 21 days 1.3 mg/m2 Velcade daily on days 1, 4, 8 and 11 20 mg dexamethasone daily on Days 1, 2, 4, 5, 8, 9, 11, 12* and 30 mg/m2 Doxil daily on day 4
Time Frame: 1 month post treatment
Population: A total of 74 patients were enrolled in this phase 1/2 study: 42 in phase 1.
Measure: Number; unit: mg
Arm/Group | Combination Drug Therapy
Number analyzed (Participants) | 42
mg
  Revlimid | 25
  VELCADE | 1.3
  Dexamethasone | 20
  Doxil | 30

2. Secondary Outcome: The Percentage of Patients That Achieved Partial or Complete Response to Treatment.
Description: Partial Response:
  * 50% reduction in the level of serum monoclonal protein for at least two determinations six weeks apart.
  * If present, reduction in 24-hour urinary light chain excretion by either, greater than or equal to 90%, or to <200 mg for at least two determinations six weeks apart.
  * 50% reduction in the size of soft tissue plasmacytomas (by clinical or radiographic examination) for at least six weeks.
  * No increase in size or number of lytic bone lesions (development of compression fracture does not exclude response).
  Complete Response:
  * Disappearance of the original monoclonal protein from the blood and urine on at least two determinations for a minimum of six weeks.
  * <5% plasma cells in the bone marrow on at least two determinations for a minimum of six weeks.
  * No increase in the size or number of lytic bone lesions.
Time Frame: 24 weeks (8, 21-day cycles)
Population: 74 patients were enrolled, but 2 were not evaluable for dose limiting toxicities. 72 patients were included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Combination Drug Therapy
Number analyzed (Participants) | 72
percentage of patients | 96

ADVERSE EVENTS:
Description: Adverse events were captured collectively for the study, not by arm, because both arms received the same drugs.
Arm/Group | Combination Drug Therapy
Serious Adverse Events (participants affected / at risk) | 3/74
Other Adverse Events (participants affected / at risk) | 24/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Drug Therapy (N=74)
Lung Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia with Grade 3 or 4 Neutropenia (Infections and infestations) | 1 (1)
Pneumonia with Normal Absolute Neutrophil Count (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Drug Therapy (N=74)
Anemia (Blood and lymphatic system disorders) | 10 (22)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (11)
Lymphopenia (Blood and lymphatic system disorders) | 5 (12)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (5)
Platelets (Blood and lymphatic system disorders) | 6 (12)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 17 (32)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 10 (14)
Diarrhea (Gastrointestinal disorders) | 6 (12)
Nausea (Gastrointestinal disorders) | 10 (11)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4 (6)
Edema: limb (General disorders) | 6 (6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 6 (9)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 (12)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (8)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (9)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (6)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5)
Dizziness (Nervous system disorders) | 7 (7)
Mood alteration (Nervous system disorders) | 5 (5)
Neuropathy: sensory (Nervous system disorders) | 7 (15)
Pain (Nervous system disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes